CLINICAL TRIAL: NCT06687226
Title: Digestion and Transit of Food DNA Through the Human Gut
Brief Title: Food DNA Digestion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00115407
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Digestion Rate
Keywords: Food; DNA; gut microbiome; transit time; digestion; digestive system; food DNA digestion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stool samples + consumption of powdered food (Other): Each participant will submit a baseline stool sample, consume a single dose of a study-specific powdered food (reconstituted in water) differing from their usual diet, and provide the subsequent five stool samples. If five samples are collected in fewer than five days, an additional sample will be obtained on the fifth day post-consumption
  Interventions: Dietary Supplement: Reconstitutable food powder

INTERVENTIONS:
Dietary Supplement: Reconstitutable food powder — During the intervention week, participants will be asked take one dose of a reconstitutable food powder provided in a ziplock bag. This powder will be a mix of Gatorade Zero Powder (1 serving) and 1 serving of commercially available powders of either one or all of the following: camu camu, kelp or maqui. The powder mix in the bag will be added to water and drunk by the participant as soon as possible after having a bowel movement (baseline stool sample). Food powders are sourced from reputable companies and are safe for consumption (Gatorade is a wellrecognized brand and available in grocery stores nationally, Navitas Organics provides certified organic, third-party tested plant food powders with fairtrade certification).

SUMMARY:
This pilot study investigates the digestion rate of naturally occurring food DNA through the human digestive tract by detecting residual food DNA in stool samples. The investigators hypothesize that food DNA primarily transits through the digestive system within 24 hours, with maximal detection in stool samples collected the day after ingestion. Previous research has focused on food DNA digestion in human gastric juices, leaving digestion through the entire gut largely unexplored. This study employs a fixed-order within subjects design involving healthy participants. Each participant will submit a baseline stool sample, consume a single dose of a study-specific powdered food (reconstituted in water) differing from their usual diet, and provide the subsequent five stool samples. If five samples are collected in fewer than five days, an additional sample will be obtained on the fifth day post-consumption. The presence and decline of food specific DNA in these samples will be quantified using qPCR, enabling us to determine the digestion rate of food DNA. The study design poses with minimal risk as it non-invasively monitors the natural process of food DNA digestion and transit through stool sample analysis.

DETAILED DESCRIPTION:
Transit time, the duration for ingested food to travel from ingestion to excretion, is crucial because it influences nutrient absorption, digestion efficiency, gut microbiome composition and the overall health of the gastrointestinal system. While numerous studies have focused on the breakdown of food components such as protein, fat and carbohydrates, the fate of food DNA, an integral part of the cells constituting these foods, remains less explored. Mouse studies indicate that food DNA can be traced in various sections of the digestive tract, with the greatest amount of degradation seen in the stomach. Human studies have supported these reports through showing significant dietary DNA degradation in the stomach and other food components in the stomach not significantly impact the efficiency of this degradation. However, this process is not 100% efficient as residual DNA has been shown to be detectable in stool in levels that are informative for health and epidemiological purposes. How long this residual DNA remains in the digestive tract and as such, the overall transit time and digestion rate for food DNA to be completely depleted from the digestive tract remain an open question.

In this study, the investigators will carry out a behavioral intervention in healthy human participants designed to investigate the transit time of dietary DNA. The design of this study is informed by the PI's previous experience with dietary interventions in human cohorts to better understand the human gut microbiome. This prior experience includes conducting a longitudinal study where samples as well as behavioral and dietary metadata were collected from human volunteers in addition to interventional studies of dietary supplements or fully controlled diets.

ELIGIBILITY:
Inclusion Criteria:

* Above age 18?
* Able to provide stool samples at no risk to the participant?
* Does the participant have card access to the MSRBIII building, and is the participant able to visit this building (at times of the participant's convenience) for the purposes of this study?

Exclusion Criteria:

* Already consume camu camu, maqui or kelp in typical diet?
* Have a history or current diagnosis of irritable bowel syndrome?
* Have a history or current diagnosis of inflammatory bowel disease?
* Have a history or current diagnosis of type 2 diabetes?
* Have a history or current diagnosis of chronic kidney disease with decreased kidney function?
* Have a history or current diagnosis of intestinal obstruction?
* Have a history or current diagnosis of untreated colorectal cancer?
* Has the participant had a colonoscopy within the past month?

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Transit time of naturally occurring food DNA through the human digestive tract | Approximately 5-8 days
  Determined by quantifying the presence of food DNA in stool samples over a specified period post-consumption.

SECONDARY OUTCOMES:
Rate of food DNA depletion | Approximately 5-8 days
  Evaluating the potential implications of the rate of food DNA depletion for nutrient absorption and gut microbiome interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence David, Principal Investigator — Duke University
Locations (1):
- Medical Sciences Research Building III (MSRB III), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No